CLINICAL TRIAL: NCT05125445
Title: Evaluation of Stability and Crestal Bone Changes Around Implants Placed at Crestal Versus Subcrestal Level in Controlled Type Two Diabetic Patients (Randomized Clinical Trial)
Brief Title: Stability and Crestal Bone Changes Around Implants Placed at Crestal Versus Subcrestal Level in Controlled Type Two Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Implants_diabetes
Record Dates: First submitted 2021-11-07; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Dental Implant; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crestally positioned implants (Experimental)
  Interventions: Procedure: Implants placed at bone crest
- Subcrestally positioned implants (Active Comparator)
  Interventions: Procedure: Implants placed 1mm Subcrestally

INTERVENTIONS:
Procedure: Implants placed at bone crest — Mid crestal incision will be performed and full-thickness envelope flap will be elevated to expose the alveolar ridge (no releasing incisions will be made).
  Implant site will be prepared according to the manufacturer's instructions under sterile copious irrigation Implants will be placed at crestal level
  Arms: Crestally positioned implants
Procedure: Implants placed 1mm Subcrestally — Implants will be placed 1mm subcrestally
  Arms: Subcrestally positioned implants

SUMMARY:
The objective of this study is to assess clinically the peri implant tissues, the radiological marginal bone loss and the stability around implants placed at the crestal versus the subcrestal level in type 2 controlled diabetic patients using cone beam computed tomography

ELIGIBILITY:
Inclusion criteria

* Type 2 controlled diabetic patients
* Patients with at least one missing tooth in lower jaw.
* Patients with sufficient alveolar ridge height and width (no need for bone augmentation).
* Patients with sufficient inter-occlusal distance that will allow future restoration.
* Patients with healthy periodontium.

Exclusion criteria

* Smokers.
* Para functional habits.
* Bad oral hygiene measured according to O'Leary plaque index.
* Pregnant women.
* Other local or systemic diseases that may compromise the surgical procedure, healing or osteointegration.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
change in Implant stability | at baseline and 3 months
  Implant stability will be measured again by Osstell at 3 different directions (buccal, mesial and distal) at the time of implant loading (after 3 months from implant placement).
change in margianl bone level | at baseline, 3rd and 6th months
  CBCT will be done Marginal bone loss in all aspects (mesial, distal buccal and lingual) The difference in distance from bone crest to apical end of the implant will be assessed at each follow up period then the mean will be calculated for mesial and distal and also for buccal and lingual.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt